CLINICAL TRIAL: NCT00873626
Title: Randomized Controled Multicentric Trial, of Non Inferiority, Comparing Two Durations of Antibiotherapy (5 Days Versus 10 Days) in COMMUNAUTARY Acute Uncomplicated Pyelonephritis.
Brief Title: Treatment's Duration of Acute Uncomplicated Pyelonephritis
Acronym: DTP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P071208
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2011-06

CONDITIONS: Urinary Tract Infection; Fever
Keywords: Urinary tract infection; treatment duration; acute pyelonephritis; good use of antibiotics
MeSH Terms: conditions — Urinary Tract Infections; Fever | interventions — Levofloxacin; Ciprofloxacin; Ofloxacin; Fluoroquinolones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): fluoroquinolones 5 days
  Interventions: Drug: levofloxacin, ciprofloxacin and ofloxacin (fluoroquinolones)
- 2 (Active Comparator): fluoroquinolones 10 days
  Interventions: Drug: levofloxacin, ciprofloxacin and ofloxacin (fluoroquinolones)

INTERVENTIONS:
Drug: levofloxacin, ciprofloxacin and ofloxacin (fluoroquinolones) — Levofloxacin 500mg : 1/j Ofloxacin : 200mgX2/j Ciprofloxacin 500mg X2/j
  Other Names: randomised duration therapy

SUMMARY:
The purpose of this study is to compare the efficacy of 5 days versus 10 days treatment duration in uncomplicated acute pyelonephritis.

Acute pyelonephritis is a common disease and the treatment duration is not found on scientific evidence. If a short treatment is equal to standard duration, it will possible to shortening antibiotherapy with ecologic and economic advantage.

DETAILED DESCRIPTION:
1. State of the issue and objective of the research The acute pyelonephritis (AP) represent the most frequent COMMUNAUTARY bacterial infection. Currently, usual recommended duration of antibiotherapy for this disease is from 10 to 21 days. The duration of treatment is not based on scientific evidence. Shortening duration of antibiotherapy would improve patient's life quality of and compliance and reduce side effects, duration of hospitalization, cost of treatment and probably limit bacterial resistance.

   The main objective of this study is to compare the rates of clinical and microbiological cure at 30 ± 5 days after the end of antibiotherapy in uncomplicated AP of young women, according to the duration of antibiotic treatment: 5 days versus 10 days.
2. People involved Patients with uncomplicated AP, will be offered to participate to the study after consultation in emergency room service or health service, in absence of non-inclusion criteria (immunodepression known, severe sepsis, allergy to antibiotics, pregnancy, lactation ...). In presence of abscesses, obstruction on the urinary tract, or infection on stranger material device requiring, in most cases, a medical-surgical treatment, they will not be eligible under the study.
3. Methods of observation or investigation restraint Non-inferiority multicenter trial, randomized in 2 parallel groups evaluating antibiotic treatment (5d vs 10d) in the uncomplicated AP.

   Recruitment and follow-up: The management of the patient will initially be provided by emergency room department or the hospital clinic. After signing the consent and inclusion (J0), the patient will receive an initial assessment, the initiation of antibiotic therapy and care. Then it will be:
   * Either in a hospital service who will follow.
   * Either by ambulatory monitoring and regularly contacted (phone with voice server) to ensure proper development.

   Randomisation will take place in J0. Finally, in all cases, a final visit will be set at J30 ± 5Day.
4. Origin and nature of the data collected - Reasons for them Data for the study duration of treatment of pyelonephritis are from information provided by patients. The nature of the data include: name, surname, date of birth, medical data (medical history, history of the disease, symptoms of infection) and telephone numbers of the patient. The collection of these numbers is essential for monitoring the patient.
5. Method for data flow These data will be confidential and only, the physician investigator, the scientific coordinator doctor, the doctor treating the patient and the clinical research fellow, will have access to this information. These data will be computerized and protected by a personal access code.
6. Duration and modalities of the research The duration of the research will be a maximum of 24 months (the duration is 12 months for inclusion and follow-up of 310 patients).

Research will multicenter (26 centers at most) and led by principal investigator (Pr. Louis Bernard) and the scientific coordinator (Dr. AURELIEN DINH) At the end of the study, all data will be destroyed.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 to 65 years old
* Non-immunocompromised
* Conducting a medical examination prior
* Signature of informed consent in writing.
* Clinical signs of urinary tract infection (urinary burning, urgency, pollakiuria, dysuria, pyuria, lumbar or pelvic pain),
* A temperature> 38 ° C,
* A positive ECBU direct seed (s) sensitive (s) to the fluoroquinolones

Exclusion Criteria:

* Antibiotic therapy prior
* Presence of complications of PNA (abscesses, dilated excretory pathways, probe urinary bladder, neurological, transplant, kidney single functional or anatomical),
* An episode of PNA within 6 months,
* having fluoroquinolones in 6 months,
* Infection on urinary endo-material (prosthetic urethral, ureteral probe)
* The immunodepressed (known seropositivity for HIV, asplenia, diabetes neutropenia, agammaglobulinemia ...)
* Pregnancy and lactation,
* Allergy to antibiotics,
* Corticosteroids concomitantly taking fluoroquinolones,
* History of TENDINOPATHY with a fluoroquinolone
* History of epilepsy
* Deficit known as glucose-6-phosphate dehydrogenase
* Life expectancy <1 month
* Cognitive major
* Patient under guardianship, CURATORSHIP or without coverage,
* The need for immunosuppressive or corticosteroid therapy,
* The need for other concomitant antibiotic treatment, whatever the cause
* No affiliation to a social security scheme (beneficiary or beneficiary).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2009-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Compare the rates of clinical and microbiological cure at 30 ± 5 days of the end of antibiotherapy in acute uncomplicated pyelonephritis of young women, according to the duration of antibiotherapy: 5 days versus 10 days. | 35 DAYS

SECONDARY OUTCOMES:
Evaluate the effectiveness bacteriological (ECBU negative direct examination and culture) of treatment to 30 ± 5 days of the end of antibiotherapy | 35 DAYS
Evaluate the clinical effectiveness of treatment: apyrexia and disappearance of clinical signs initial J2 ± 1; J5 ± 1, ± 1 of J10 beginning of treatment and 30 ± 5 days of the end of antibiotherapy, | 35 DAYS
Identifying risk factors for failure of antibiotic treatment (co-morbidities, bacteremia) | 35 DAYS
Assessing the tolerance of the antibiotic, the presence of adverse events related to drug | 35 DAYS
To assess adherence to treatment, the proportion of patients observant good, average and low observant | 35 DAYS
Assess the changes in sensitivity to antibiotics (fluoroquinolones) in the nasal flora, pharyngeal and digestive. | 35 DAYS

CONTACTS AND LOCATIONS:
Overall Officials: Louis BERNARD, MD PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (2):
- France (2):
  - University hospital of Garches, Garches
  - university hospital of TOURS, Tours